CLINICAL TRIAL: NCT02987218
Title: Comparison Of Pharmacological Neuroprotection Provided By PROPOFOL VERSUS DESFLURANE For Long Term Postoperative Cognitive Dysfunction In Patients Undergoing Surgery For Aneurysmal Subarachnoid Hemorrhage
Brief Title: Comparison of Neuroprotection by Propofol and Desflurane for POCD Following Subarachnoid Hemorrhage Surgery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Dr Shalvi mahajan, Senior Resident, Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: INT/IEC/2015/741
Record Dates: First submitted 2016-11-13; First posted 2016-12-08 (Estimated); Last update posted 2016-12-08 (Estimated); Status verified 2016-12

CONDITIONS: Postoperative Cognitive Function
Keywords: POCD; subarachnoid hemorrhage; Propofol; Desflurane
MeSH Terms: conditions — Subarachnoid Hemorrhage | interventions — Propofol; Desflurane

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- PROPOFOL (Active Comparator): Intravenous hypnotic agent Decrease Cerebral Metabolic reduction Decrease ICP(Intracranial pressure) Better cognitive Function preservation
  Interventions: Drug: Propofol
- DESFLURANE (Active Comparator): Inhalational agent. Decreases cerebral metabolism Increase /decreases ICP Cognition preservation
  Interventions: Drug: Desflurane

INTERVENTIONS:
Drug: Propofol — Intravenous hypnotic agent Decrease Cerebral Metabolic reduction Decrease ICP Better cognitive Function preservation
  Arms: PROPOFOL
Drug: Desflurane — Inhalational agent. Decreases cerebral metabolism Increase /decreases ICP Cognition preservation
  Arms: DESFLURANE

SUMMARY:
Aneurysmal subarachnoid hemorrhage (aSAH) is characterized by the rupture of an intracranial aneurysm and accumulation of blood in the subarachnoid space with 30 to 40% mortality rate. Amongst the survivors 40-50% suffers disability due to cognitive decline.Trends towards early surgery offers challenge to anesthesiologist to provide optimum brain relaxation and simultaneously maintaining stable hemodynamics. Anesthetic agents are administered to conduct smooth neurosurgical procedure. These agents may affect patient's cognitive function postoperatively.Currently most common anesthetic agents used are either intravenous hypnotic agents (propofol) or volatile inhalational agents (isoflurane/sevoflurane/desflurane). Provision of neuroprotection with propofol and volatile inhalational agents has been studied by various authors.Not many studies have been performed in patients undergoing aneurysmal clipping surgeries looking into effects of various anesthetic agents on intraoperative (I/O) brain condition, I/O hemodynamic and POCD.Thus present study is planned to compare propofol and desflurane for long term postoperative cognitive decline in patients undergoing surgery following aneurysmal subarachnoid hemorrhage.

DETAILED DESCRIPTION:
100 patients will be randomized into two groups, Desflurane group (Group D) and Propofol group (Group P) using a computer generated algorithm. Written informed consent will be taken from all the patients.

Cognition assessed using MOCA (Montreal Cognitive Assessment)test. A preoperative assessment for establishing the patient's baseline performance. Surgery-related factors may affect test performance if performed too early to reduce possibility of confounding factors, we planned to conduct the test for POCD at the time of discharge of the patient after surgery. To compare long term protection provided by anesthetic agent cognitive functions were assessed at one month following surgery.

Cognitive functions will be assessed at following time period A) Preoperatively B) Postoperatively B1- At the time of discharge B2- 1month after discharge following surgery.

Biomarker levels S100B levels were also measured A) Preoperatively B) Intraoperatively - post clipping C) Postoperatively - 1hour after surgery

ELIGIBILITY:
Inclusion Criteria:

1. Patients scheduled for aneurysmal SAH surgery with clinical and radiological evidence of cerebral aneurysm.
2. Age between 18 to 65 yrs.
3. World Federation of neurosurgery grade 1, 2.
4. American society of Anesthesia grade 1, 2 and 3.

Exclusion Criteria:

1. Co-morbidities other than hypertension and diabetes mellitus like cardiovascular disease and respiratory impairment.
2. Patients with known psychiatric disease.
3. History of drug abuse.
4. Low level of education (illiterate) or multiple failures in school.
5. Patients who are unconscious, intubated or tracheostomised even after two weeks following exposure to anesthesia will also be excluded from the study.
6. Intraoperative complications like massive blood loss, prolonged clipping time(>20minutes), severe intraoperative brain swelling precluding replacement of bone flap.
7. Patients with infectious diseases and respiratory complications.
8. Multiple surgeries.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2015-07; Primary Completion 2016-10 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Assessment of cognitive function at one month following surgery. | One month
  Montreal Cognitive Assessment scale is used

SECONDARY OUTCOMES:
Assessment of cognitive function preoperatively Assessment of cognitive function at discharge. Comparison of biomarker of cognitive dysfunction | Baseline cognition assessment prior to surgery
  Montreal Cognitive Assessment scale used
Assessment of cognitive function preoperatively Assessment of cognitive function at the time of discharge from hospital | Discharge from hospital
  Montreal Cognitive Assessment scale used
Comparison of biomarker (S-100B) levels | Prior to surgery , After clipping of aneurysm, One hour after completion of surgery
  Blood sample for S100B levels used

CONTACTS AND LOCATIONS:
Overall Officials: Shalvi Mahajan, MD, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh; Hemant Bhagat, DM, Principal Investigator — Post Graduate Institute of Medical Education and Research, Chandigarh
Locations (1):
- Postgraduate institute of medical education and research, Chandigarh, Chandigarh, India

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Result] Wong GK, Lam S, Ngai K, Wong A, Mok V, Poon WS; Cognitive Dysfunction after Aneurysmal Subarachnoid Haemorrhage Investigators. Evaluation of cognitive impairment by the Montreal cognitive assessment in patients with aneurysmal subarachnoid haemorrhage: prevalence, risk factors and correlations with 3 month outcomes. J Neurol Neurosurg Psychiatry. 2012 Nov;83(11):1112-7. doi: 10.1136/jnnp-2012-302217. Epub 2012 Jul 31. PMID 22851612